CLINICAL TRIAL: NCT03825627
Title: From Attention to Behavior: Increasing Behavioral Inhibition Through Transcranial Direct Current Stimulation in Pedophilia
Brief Title: From Attention to Behavior: Increasing Behavioral Inhibition
Acronym: tDCS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018-02028
Record Dates: First submitted 2019-01-22; First posted 2019-01-31 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Pedophilia
MeSH Terms: conditions — Pedophilia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Antisaccade Task (active tDCS) (Active Comparator): During the antisaccade task, the investigators will show participants computer-generated images depicting clothed and sexually relevant (nude) children, young adults and adults of both genders. Images will be drawn from the Virtual People Set and the Not-Real-People Set (Pacific Psychological Assessment Corporation, 2004). Pedophilic participants are expected to show a sexual preference towards a prepubescent body scheme whereas stimuli displaying adolescence and adulthood (sexual maturity) are expected to be sexually preferred by the teleiophilic control participants. In this arm active Transcranial Direct Current Stimulation will be used to influence performance.
  Interventions: Device: Transcranial Direct Current Stimulation
- Antisaccade Task (sham tDCS) (Sham Comparator): During the antisaccade task, the investigators will show participants computer-generated images depicting clothed and sexually relevant (nude) children, young adults and adults of both genders. Images will be drawn from the Virtual People Set and the Not-Real-People Set (Pacific Psychological Assessment Corporation, 2004). Pedophilic participants are expected to show a sexual preference towards a prepubescent body scheme whereas stimuli displaying adolescence and adulthood (sexual maturity) are expected to be sexually preferred by the teleiophilic control participants. In this arm sham Transcranial Direct Current Stimulation will be used during the task.
  Interventions: Device: Transcranial Direct Current Stimulation
- Approach Avoidance Task (active tDCS) (Active Comparator): During the Approach-Avoidance Task (AAT), participants will look at a series of images depicting children and adults wearing swimsuits. The images were sampled from internet advertisements and do not constitute legally objectionable material. When sourcing the images, rigorous attention was paid to meet the criteria for fair use indicated by the American Psychological Association. There are 160 images in total. Half of the images will be used in the active and the other half in the sham condition (i.e., 20 female adults, 20 female children, 20 male adults, and 20 male children per condition). In this arm active Transcranial Direct Current Stimulation will be used to influence performance.
  Interventions: Device: Transcranial Direct Current Stimulation
- Approach Avoidance Task (sham tDCS) (Sham Comparator): During the Approach-Avoidance Task (AAT), participants will look at a series of images depicting children and adults wearing swimsuits. The images were sampled from internet advertisements and do not constitute legally objectionable material. When sourcing the images, rigorous attention was paid to meet the criteria for fair use indicated by the American Psychological Association. There are 160 images in total. Half of the images will be used in the active and the other half in the sham condition (i.e., 20 female adults, 20 female children, 20 male adults, and 20 male children per condition). In this arm sham Transcranial Direct Current Stimulation will be used during the task.
  Interventions: Device: Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — Conductive saline-soaked rubber electrodes super-imposed on sponge plates will be placed on the scalp at F3 (active electrode, 4.4×4.4cm) and on the contralateral supraorbital area (reference electrode, 5.1×10.2cm).
  Stimulation will be applied using a battery-driven constant-current regulator (Oasis Pro, Edmonton, Alberta, Canada). For each stimulation, the direct current is initially increased in a ramp-like fashion over 10 s until reaching 2 milliampere (mA) and will be similarly decreased at the end of stimulation.
  In the active tDCS condition, stimulation will be maintained for 20 min; in the sham condition, it will be turned off after 15 s of stimulation, with a ramp-up/down of 10 s (i.e., 35 s total).

SUMMARY:
This project will investigate if transcranial direct current stimulation can be used as treatment for Pedophilia. Treatment efficacy will be evaluated with behavioral tasks and the recording of eye-movement.

DETAILED DESCRIPTION:
Pedophilia is an important motivation for sexual offenses involving children, including child pornography and sexual contacts with children (henceforth, pedosexual behavior). Indeed, approximately half of individuals convicted for sexual offenses against children have a Pedophilic disorder and offenders with a Pedophilic disorder are much more likely to sexually reoffend.

A promising line of research has examined the neurocognitive basis of pedophilia. Pedophilic individuals display altered activity in the dorsolateral prefrontal cortex (dlPFC) when attending to child-related stimuli. This brain area is involved in the cognitive control of sexual arousal. Transcranial Direct Current Stimulation (tDCS) has been examined as a non-invasive method to increase activity in the dlPCF, ultimately increasing inhibitory control over impulses. Accumulating evidence also shows that individuals have an attentional bias towards sexually preferred stimuli. These attentional processes can be investigated by recording eye movements. Early automatic eye movements are particularly relevant in discriminating individuals with pedophilia from those without pedophilia.

The proposed study will examine the effects of tDCS over the dlPFC of pedophilic individuals and healthy controls, while they complete a task requiring controlled attention to virtual (computer-generated) images of children and adults. In two separate sessions, participants will be randomly assigned to an active and a placebo (sham) tDCS condition. Eye movements will be recorded during the task.

The investigators expect to observe a conflict between automatic and controlled attention when participants are presented with their sexually preferred stimuli. Specifically, the investigators expect pedophiles to show an attentional bias towards virtual child stimuli. The investigators predict that the attentional conflict will be reduced when tDCS is applied, compared to the sham condition. If the attentional bias is a key cognitive feature of sexual interest, the investigators expect to measure changes in reported or indirectly assessed sexual preferences.

ELIGIBILITY:
Inclusion Criteria:

Patients

* Diagnosed with pedophilia (further psychiatric illnesses possible)
* Sufficient German language skills

Controls:

* Not diagnosed with Pedophilia (or other psychiatric illnesses)
* Sufficient German language skills

Exclusion Criteria:

Patients

* Prior head injury with loss of consciousness for at least 5 min
* Neurological diagnosis (including epilepsy) or prior medical conditions with possible central nervous system sequelae
* Metallic implants inside the brain or any electrical medical device (e.g. pacemaker) in the body
* Visual or hearing impairment, to the extent that it interferes with task instructions

Current medication in patients (antiandrogenic medication among the pedophilic subjects, in particular) will be recorded and acknowledged as a covariate.

Controls

* Prior head injury with loss of consciousness for at least 5 min
* Neurological diagnosis (including epilepsy) or prior medical conditions with possible central nervous system sequelae
* Metallic implants inside the brain or any electrical medical device (e.g. pacemaker) in the body
* Visual or hearing impairment, to the extent that it interferes with task instructions
* Current or previous pedophilic sexual interest

For both groups further exclusion (prematurely) will occur if initial data shows that participants don't comply with instructions or if questionnaires hint toward a lack of sexual interest in general.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Entry Time | Through study completion, an average of 10 months. The outcome measure is not an event but a performance measure recorded for every participant in every session.
  In the Antisaccade task entry time will be recorded with an eye-tracker in both active and sham tDCS conditions. Time to first fixation (entry time) is defined as the time from stimulus onset to the first fixation directed to the target stimulus. This index can be treated as reaction time (RT) and will provide a measure of controlled attention. The location of the first fixation indicates which stimulus captures subject's automatic attention. The proportion of correct/incorrect fixations (%) will inform us about automatic attentional processes. Thus entry time is a single performance index measured with a unit of time, in this case Milliseconds (ms). Every participant's performance in the Antisaccade task will be measured with entry time (ms) as well as the percentage (%) of correct responses. Since the task is not difficult, the percentage values only serve to check for compliance with task instructions. The real focus of the study lies in the RT as recorded with entry time in ms.
differential AAT index (∆RT) | Through study completion, an average of 10 months. The outcome measure is not an event but a performance measure recorded for every participant in every session.
  In the Approach-Avoidance Task (AAT) the differential AAT index (∆RT) will be recorded in both active and sham tDCS condition using the response on the joystick. The proportion of correct/incorrect responses (%) will inform us about automatic attentional processes. Thus the ∆RT is a single performance index for speed tests measured with a unit of time, in this case Milliseconds (ms). It gives information on how fast participants responded using the joystick. In addition, the percentage (%) of correct responses with the joystick will be recorded. Since the task is not difficult, the percentage values only serve to check for compliance and if task instructions were understood. The real focus of the study lies in the RT as recorded with ∆RT in ms.

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Brackmann, Dr., Principal Investigator — University Hospital of Psychiatry Zurich, Department of Forensic Psychiatry
Locations (1):
- Psychiatrische Universitätsklinik Zürich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dombert B, Mokros A, Bruckner E, Schlegl V, Antfolk J, Backstrom A, Zappala A, Osterheider M, Santtila P. The virtual people set: developing computer-generated stimuli for the assessment of pedophilic sexual interest. Sex Abuse. 2013 Dec;25(6):557-82. doi: 10.1177/1079063212469062. Epub 2013 Jan 7. PMID 23296092
- [Background] Cacioppo JT, Priester JR, Berntson GG. Rudimentary determinants of attitudes. II: Arm flexion and extension have differential effects on attitudes. J Pers Soc Psychol. 1993 Jul;65(1):5-17. doi: 10.1037//0022-3514.65.1.5. PMID 8355142
- [Background] Ettinger U, Ffytche DH, Kumari V, Kathmann N, Reuter B, Zelaya F, Williams SC. Decomposing the neural correlates of antisaccade eye movements using event-related FMRI. Cereb Cortex. 2008 May;18(5):1148-59. doi: 10.1093/cercor/bhm147. Epub 2007 Aug 28. PMID 17728263
- [Background] Fromberger P, Jordan K, Steinkrauss H, von Herder J, Witzel J, Stolpmann G, Kroner-Herwig B, Muller JL. Diagnostic accuracy of eye movements in assessing pedophilia. J Sex Med. 2012 Jul;9(7):1868-82. doi: 10.1111/j.1743-6109.2012.02754.x. Epub 2012 Apr 30. PMID 22548761
- [Background] Oberlader VA, Ettinger U, Banse R, Schmidt AF. Development of a Cued Pro- and Antisaccade Paradigm: An Indirect Measure to Explore Automatic Components of Sexual Interest. Arch Sex Behav. 2017 Nov;46(8):2377-2388. doi: 10.1007/s10508-016-0839-7. Epub 2016 Oct 17. PMID 27752855
- [Background] Phaf RH, Mohr SE, Rotteveel M, Wicherts JM. Approach, avoidance, and affect: a meta-analysis of approach-avoidance tendencies in manual reaction time tasks. Front Psychol. 2014 May 8;5:378. doi: 10.3389/fpsyg.2014.00378. eCollection 2014. PMID 24847292
- [Background] Poeppl TB, Nitschke J, Santtila P, Schecklmann M, Langguth B, Greenlee MW, Osterheider M, Mokros A. Association between brain structure and phenotypic characteristics in pedophilia. J Psychiatr Res. 2013 May;47(5):678-85. doi: 10.1016/j.jpsychires.2013.01.003. Epub 2013 Feb 9. PMID 23399486
- [Background] Weidacker K, Kargel C, Massau C, Weiss S, Kneer J, Krueger THC, Schiffer B. Approach and Avoidance Tendencies Toward Picture Stimuli of (Pre-)Pubescent Children and Adults: An Investigation in Pedophilic and Nonpedophilic Samples. Sex Abuse. 2018 Oct;30(7):781-802. doi: 10.1177/1079063217697134. Epub 2017 Mar 20. PMID 29188755